CLINICAL TRIAL: NCT02739646
Title: The Representation of the Sensibility of the Breast on the Somatosensory Cortex Using 7 Tesla fMRI: A Pilot Study
Brief Title: The Representation of the Sensibility of the Breast on the Somatosensory Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Rene van der Hulst, Prof. dr., Maastricht University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NL54890.068.15
Record Dates: First submitted 2016-04-06; First posted 2016-04-15 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Healthy
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Females (Experimental): Functional MRI scan of the somatosensory cortex while the breast skin is stimulated by piezo-stimulators.
  Interventions: Device: Functional MRI scan
- Males (Experimental): Functional MRI scan of the somatosensory cortex while the breast skin is stimulated by piezo-stimulators.
  Interventions: Device: Functional MRI scan

INTERVENTIONS:
Device: Functional MRI scan — 7.0 Tesla functional MRI scan

SUMMARY:
Rationale: The representation of the breast on the somatosensory cortex has not been precisely located. Therefore, a pilot study with healthy subjects is needed to localize the sensibility of the breast on the somatosensory cortex with the use of a 7 Tesla fMRI.

Objective: To determine the exact localization of the representation of the sensibility of the breast and nipple-areola complex on the somatosensory cortex. Secondly, to assess whether there are differences in representation between individuals of the same sex and between both sexes.

Study design: A single center pilot study carried out in the Maastricht University Medical Center, the Netherlands.

Study population: A total of 10 female and 10 male healthy individuals will be recruited.

Intervention: Every subject will undergo a functional MRI scan with stimulators applied to the bare breast in a fixed pattern. These stimulate the skin and sensory nerves of the breast and nipple-areola complex in a random sequence.

Main study parameters: The hemodynamic response after stimulation of the skin of the breast and nipple-areola complex, representing neuronal activity in that region, is measured. Within the somatosensory cortex (S1 and S2), the temporo-spatial brain activity patterns after the various stimulation conditions are assessed, and the representation of the breast on the somatosensory cortex is mapped.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Between 21 and 35 years old
* Healthy; i.e. no comorbidities
* Women: breast size cup B or C
* BMI < 27.0 kg/m2
* Informed consent

Exclusion Criteria:

* Any comorbidities
* Previous breast operation of any kind
* Previous allergic reactions to adhesives or plasters
* Any MRI exclusion criteria e.g.:

(No piercings or other iron materials (except a metal brace behind front teeth) (Claustrophobia)

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-13; Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Changes in the blood oxygen level dependent (BOLD) contrast as a function of vibrotactile stimulation of the breast and nipple-areola complex | 90 minutes
  Changes will be analysed using multi-voxel pattern analysis to localize the different parts of the breast in the somatosensory cortex.

SECONDARY OUTCOMES:
Changes in the blood oxygen level dependent (BOLD) contrast as a function of vibrotactile stimulation of the breast and nipple-areola complex in males compared to females | 90 minutes
  Differences between both sexes in localization or representation of the breast in the somatosensory cortex will be assessed.
Changes in the blood oxygen level dependent (BOLD) contrast as a function of vibrotactile stimulation of the breast and nipple-areola complex between individuals of the same sex | 90 minutes
  Differences between individuals of the same sex in localization or representation of the breast in the somatosensory cortex will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Rene van der Hulst, prof,MD,PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided